CLINICAL TRIAL: NCT03884244
Title: The Effect of Postoperative Chewing Gum on Intestinal Functions After Gynecological Laparoscopic Surgery
Brief Title: Postoperative Chewing Gum and Gynecological Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, principal investigator, M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018.10.21
Record Dates: First submitted 2019-03-12; First posted 2019-03-21 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Gynecologic Disease; Postoperative Ileus; Paralytic Ileus
Keywords: Laparoscopic Surgery; Postoperative Bowel Function
MeSH Terms: conditions — Genital Diseases, Female; Intestinal Pseudo-Obstruction | interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- taking chewing gum patients (Active Comparator)
  Interventions: Other: chewing gum
- no chewing gum (No Intervention)

INTERVENTIONS:
Other: chewing gum — The group who take chewing gum after operation
  Arms: taking chewing gum patients

SUMMARY:
The authors aimed to evaluate the effects of postoperative gum chewing on laparoscopic gynecological surgery, gastrointestinal function-intestinal mobility and early postoperative recovery. Patients undergoing elective gynecological laparoscopy were randomized. Demographic and characteristic features of the patients were recorded. Operation type, operation and anesthesia information were recorded. Patients underwent a postoperative routine regimen. Starting from the sixth hour, the sugar-free gum was crushed every 15 minutes until the gas was released. Postoperative follow-up was performed routinely. The first bowel movements, first bowel movements and first gas extraction and first decongestation periods were recorded.

DETAILED DESCRIPTION:
The team of the research team of the research team will listen and record the bowel sounds of the patients, using a stethoscope every two hours starting from the postoperative 3rd hour until the first bowel sounds are heard in each patient.

Patients who were able to tolerate patients starting from the 8th hour after the surgery were allowed for mobilization. Also, they were allowed to take fluid regimen from the postoperative 12th hour. Patient satisfaction was evaluated by using visual analogue scale (VAS) on the day of discharge on chewing postoperative.

The primary index for the return of GI functions was the first gas removal time. Secondary index was the time of first bowel sound, the first time of admission, hospitalization time and the presence of postoperative ileus.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparoscopic gynecological surgery.

Exclusion Criteria:

* Those who have been operated for malignant reasons,
* Those who underwent emergency surgery,
* Who could not chew gum,
* Who had serious surgical complications (postoperative intraabdominal hemorrhage, infection, peritonitis),
* Who had a history of gastrointestinal disease,
* Secondary laparotomy.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Bowel Functions | Postoperative first 1440 minutes
  The Effect of Postoperative Chewing Gum on Intestinal Functions after Gynecological Laparoscopic Surgery ; The primary index for the return of GI functions was the first gas removal time. Patient first extraction of gas, recorded in minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Pınar Kadiroğulları, Istanbul, Turkey (Türkiye)